CLINICAL TRIAL: NCT07070908
Title: Modifications to Gastric Tube Construction in Vertical Gastrectomy: Implications for Gastroesophageal Reflux Disease and Patient Quality of Life
Brief Title: Modifications to Gastric Sleeve: Implications for GRED and Quality of Life
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Juan de Dios Tenerife (Other)
Collaborators: Hospital Regional de Malaga (Other)
Responsible Party: Principal Investigator, Julen Ramon Rodríguez, Principal Investigator, Hospital San Juan de Dios Tenerife
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 25-00101
Record Dates: First submitted 2025-06-27; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Obese Patients (BMI ≥ 30 kg/m²); Obese Patients; Obese Patients With Bariatric Surgery; Obese With Comorbidities
Keywords: Obesity; Vertical gastrectomy; Gastroesophageal reflux disease; Quality of life
MeSH Terms: conditions — Obesity; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- No antrum or fundus calibration (Experimental): No antrum or fundus calibration
  Interventions: Procedure: No antrum calibration; Procedure: No fundus calibration
- Fundus calibration (Experimental): Fundus calibration only
  Interventions: Procedure: Fudus calibration; Procedure: No antrum calibration
- Antrum and fundus calibration (Experimental): Antrum and fundus calibration
  Interventions: Device: Antrum calibration; Procedure: Fudus calibration
- Antrum calibration (Experimental): Antrum calibration only
  Interventions: Device: Antrum calibration; Procedure: No fundus calibration

INTERVENTIONS:
Device: Antrum calibration — For antral calibration, a 50 cc balloon catheter was used to guide the staple line.
  Other Names: Antrum section
  Arms: Antrum and fundus calibration; Antrum calibration
Procedure: Fudus calibration — Fundus transection was performed 1 cm from the "fat pad" in calibrated cases (an anatomically constant area near the short gastric vessels that contains minimal fat and facilitates dissection toward the diaphragmatic crus).
  Other Names: fundus section
  Arms: Antrum and fundus calibration; Fundus calibration
Procedure: No antrum calibration — In patients without antrum calibration, gastric transection was performed 5 cm from the pylorus.
  Arms: Fundus calibration; No antrum or fundus calibration
Procedure: No fundus calibration — Fundus transection was performed adjacent to the "fat pad" in no calibrated cases.
  Arms: Antrum calibration; No antrum or fundus calibration

SUMMARY:
This is a prospective randomized clinical trial evaluating the impact of antrum and fundus calibration during laparoscopic vertical gastrectomy (VG) on postoperative gastroesophageal reflux disease (GERD), quality of life, and surgical costs. Eligible participants are adults with morbid obesity (BMI ≥35 kg/m²) undergoing LSG. Patients are randomized into four groups based on whether antral and/or fundal calibration is performed. Primary outcomes include the incidence of de novo GERD at 12 months. Secondary outcomes include postoperative quality of life, vomiting , surgical complications, weight loss, and operative costs. The study aims to optimize the LSG technique by identifying anatomical modifications that minimize GERD while improving clinical outcomes

DETAILED DESCRIPTION:
This is a prospective, randomized clinical trial conducted at the Regional University Hospital of Málaga. The objective is to evaluate the effect of antrum and fundus calibration during vertical gastrectomy (VG) on the incidence of gastroesophageal reflux disease (GERD), quality of life, weight loss, and surgical costs.

Eligibility Criteria:

Inclusion criteria include adults with an indication for VG, a body mass index (BMI) ≥ 35 kg/m², and provision of written informed consent.

Exclusion criteria include endocrine-related obesity, active gastrointestinal disease (such as GERD, esophagitis, peptic ulcer, or motility disorders), or a history of gastric surgery.

Randomization and Study Arms:

Patients are randomized to one of four groups:

Group A: No antrum or fundus calibration Group B: Fundus calibration only Group C: Antrum and fundus calibration Group D: Antrum calibration only

Surgical Protocol:

All patients receive a 36 Fr bougie to shape the gastric tube. In cases with antrum calibration, a 50 cc balloon catheter (MidSleeve®) guides the staple line. For fundus calibration, transection is performed 1 cm from the anatomical fat pad. Stapler height is adjusted according to tissue thickness, and the staple line is reinforced.

GERD Assessment:

De novo GERD is defined by endoscopic findings (esophagitis), pathological pH monitoring (DeMeester index > 14.72 or acid exposure > 4%), or clinically significant reflux symptoms with a GERD-HRQL score ≥ 12. Preoperative GERD is ruled out by endoscopy and questionnaire, followed by pH monitoring if symptoms are present.

Follow-Up and Monitoring:

Patients are followed at 2 weeks, 3, 6, and 12 months. In those reporting symptoms postoperatively, endoscopy and pHmetry are repeated.

Variables Collected:

Data include age, sex, BMI, comorbidities, operative details (e.g., number of stapler cartridges), complications (Clavien-Dindo classification), weight loss (%EWL), quality of life metrics (vomiting, regurgitation, satiety, food tolerance), and presence of GERD.

Statistical Analysis:

Comparisons are made across the four study groups, as well as pooled analyses for fundus calibration (yes vs. no) and antrum calibration (yes vs. no). Quantitative data are analyzed using Student's t-test or Mann-Whitney U test, and categorical variables by chi-square or Kruskal-Wallis test as appropriate. Spearman's correlation is used for association between variables. A p-value < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with morbid obesity on the waiting list for bariatric surgery.
* Both male and female participants.
* Age between 18 and 65 years.
* BMI > 35 kg/m².
* Availability to attend scheduled follow-up visits.
* Indication for sleeve gastrectomy as the first bariatric procedure.

Exclusion Criteria:

* Obesity of endocrine origin.
* Preoperative GERD (diagnosed by pH-metry or upper endoscopy following a positive GERD-HRQL test).
* Active gastrointestinal disease (such as esophagitis, peptic ulcer, cancer, or esophageal motility disorder), diagnosed by endoscopy or manometry.
* History of previous gastric surgery.
* Patients not meeting the inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-04-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of de novo Gastroesophageal Reflux Disease (GERD) | 12 months postoperatively
  De novo GERD will be diagnosed if any of the following criteria are met:
  Presence of esophagitis according to the Los Angeles classification DeMeester index > 14.72 Acid exposure time > 4% on 24-hour pH-metry GERD-HRQL questionnaire score ≥ 12

SECONDARY OUTCOMES:
Incidence of Postoperative Vomiting | 12 months postoperatively
  Postoperative vomiting will be assessed during follow-up visits at 2 weeks, 3 months, 6 months, and 12 months. Patients will self-report the presence, frequency, and severity of vomiting episodes related to food intake.
Incidence of Postoperative Regurgitation | 12 months postoperatively
  Postoperative regurgitation will be assessed during follow-up visits at 2 weeks, 3 months, 6 months, and 12 months. Patients will self-report the presence, frequency, and severity of regurgitation related to food intake. In addition, regurgitation will be evaluated using the specific item in the GERD-Health-Related Quality of Life (GERD-HRQL) questionnaire.
Food intake volume per meal | 12 months postoperatively
  Food intake volume will be assessed during follow-up visits at 2 weeks, 3 months, 6 months, and 12 months.
Percentage of excess weight loss (%EWL) | 12 months postoperatively
  The percentage of excess weight loss (%EWL) will be calculated at 12 months postoperatively. %EWL is defined as:
  Ideal weight will be based on a BMI of 25 kg/m². This measure evaluates the effectiveness of the procedure in achieving weight reduction
Change in Hypertension Status from Baseline to 12 Months Post-Surgery | Baseline and within 12 months after surgery
  Hypertension improvement or resolution will be determined by comparing preoperative and postoperative clinical records, and antihypertensive medication usage.
Postoperative BMI | Within 12 months after surgery
  The Body Mass Index (BMI) will be calculated at each postoperative follow-up visit (2 weeks, 3 months, 6 months, and 12 months) to assess the evolution of weight loss. BMI is calculated as weight in kilograms divided by the square of height in meters (kg/m²)
Weight loss | Within 12 months after surgery
  Weight loss will be calculated at each postoperative follow-up visit (2 weeks, 3 months, 6 months, and 12 months)
Postoperative Morbidity | Up to 30 days after surgery
  Postoperative complications will be assessed and classified according to the Clavien-Dindo classification system. All adverse events occurring within 30 days of surgery will be recorded and categorized by severity.
Number of stapler cartridges used | During the surgical procedure
  The total number of stapler cartridges used during vertical gastrectomy will be recorded for each patient.
Intraoperative complications | During the surgical procedure
  All adverse events occurring during surgery will be recorded, including bleeding, injury to adjacent organs, anesthetic incidents, or other unforeseen technical difficulties
Change in Type 2 Diabetes Mellitus Status from Baseline to 12 Months Post-Surgery | Baseline and within 12 months after surgery
  Improvement or resolution of Type 2 Diabetes Mellitus will be assessed through levels, HbA1c, and antidiabetic medication requirements
Change in Hypercholesterolemia Status from Baseline to 12 Months Post-Surgery | Baseline and within 12 months after surgery
  Evaluated through serum cholesterol levels and lipid-lowering medication usage before and after surgery.
Change in Obstructive Sleep Apnea Syndrome (OSAS) Status from Baseline to 12 Months Post-Surgery | Baseline and within 12 months after surgery
  Improvement or resolution based on patient-reported symptoms, CPAP usage, and clinical evaluation
Change in Hypertriglyceridemia Status from Baseline to 12 Months Post-Surgery | Baseline and within 12 months after surgery
  Improvement or resolution of hypertriglyceridemia will be assessed by comparing preoperative and postoperative triglyceride levels and the need for lipid-lowering therapy
Change in Postoperative Satiety Over Time | 2 weeks, 3 months, 6 months, and 12 months postoperatively
  Satiety will be assessed through patient self-reported feedback during postoperative visits at 2 weeks, 3 months, 6 months, and 12 months. The evaluation includes perceived fullness after meals and the volume of food tolerated per intake.
Tolerance to Oral Liquid Intake After Surgery | 2 weeks, 3 months, 6 months, and 12 months postoperatively
  Tolerance to oral liquid intake will be assessed at 2 weeks, 3 months, 6 months, and 12 months after surgery. This variable evaluates the patient's ability to ingest and retain clear liquids without nausea, vomiting, or discomfort. Data will be collected through clinical interviews, patient-reported outcomes, and medical records during scheduled follow-up visits.
Tolerance to Oral Solid Intake After Surgery | 2 weeks, 3 months, 6 months, and 12 months postoperatively
  Assessment of the patient's ability to tolerate solid food intake following vertical gastrectomy. Tolerance will be evaluated based on patient self-reported ability to consume solid foods without discomfort, vomiting, or regurgitation.
Tolerance to Oral Meat Intake After Surgery | 2 weeks, 3 months, 6 months, and 12 months postoperatively
  Patient-reported ability to consume and tolerate meat (solid protein) without nausea, vomiting, regurgitation, or abdominal discomfort. Data will be collected via clinical interviews at each postoperative visit

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Francisco Javier Moreno Ruiz, MD Head of the Bariatric Surgery Unit, Study Director — Regional University Hospital of Málaga
Locations (1):
- Regional University Hospital of Málaga, Málaga, Malaga, Spain

IPD SHARING:
Plan to Share IPD: No
The data presented in this study are available on request from the corresponding author, in accordance with the informed consent provided by study participants and subject to patient confidentiality and data protection policies